CLINICAL TRIAL: NCT05755737
Title: A Proof of Principle Study of Ondansetron for the Prevention of Vasovagal Syncope: The Eleventh Prevention of Syncope Trial (POST11)
Acronym: POST 11
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POST 11
Record Dates: First submitted 2023-02-09; First posted 2023-03-06 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Vasovagal Syncope (VVS); Syncope
Keywords: Ondansetron
MeSH Terms: conditions — Syncope, Vasovagal; Syncope | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron (Active Comparator): 2 doses of Ondansetron 8mg PO (evening before and morning of study)
  Interventions: Drug: Ondansetron
- Placebo (Active Comparator): 2 doses of matching placebo 8 mg PO (evening before and morning of study)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — Serotonin antagonists (5-HT3 antagonists) (Carbazole Derivative)
  Arms: Ondansetron
Drug: Placebo — Matching placebo identical in appearance.
  Arms: Placebo

SUMMARY:
About 20% of adults faint recurrently. These patients are often highly symptomatic, have problems with employment and driving, can be injured, and have poor quality of life. There are few therapies that have withstood the test of randomized clinical trials. the investigators will conduct a prospective, randomized, parallel, double-blind, proof-of-concept study that tests the hypothesis that serotonin 5HT3 receptor inhibition with ondansetron prevents tilt-induced vasovagal syncope (VVS) and pre-syncope in patients with clinical VVS. A total of 70 patients with quantitative clinical diagnostic criteria for VVS and at least 1 syncopal spell in the preceding year will be randomized in a double-blind acute phase 2 study to ondansetron 8 mg PO BID x 2 doses or matching placebo. The endpoint will be presyncope or syncope associated with diagnostic hemodynamic changes. These data should provide useful preliminary data as a foundation on which to conduct a subsequent randomized clinical trial.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, parallel-arm study in which the subjects will undergo a tilt table test following 2 doses of ondansetron 8 mg PO (evening before and morning of study) or after 2 doses of matching placebo (on separate days). On the morning of the study, the fasting subject (except for medications) will be instrumented, on an empty bladder. ECG electrodes will be applied to monitor continuous heart rhythm. BP will be monitored continuously using a finger volume clamp method using one or more of several extant devices, and calibrated with intermittent brachial cuff measurements. One intravenous cannula will be placed in the contralateral arm (to the BP cuff) for blood sampling.

3.9. Tilt Table Protocol: Following the insertion of the venous cannulae, a period of at least 20 minutes will be allowed to elapse before a 10-minute basal control (baseline) period. Baseline data will be digitally recorded in this time. In the last 5 minutes of this period, blood will be drawn for fractionated plasma catecholamines. The table will be rapidly raised to 80 degrees for up to 60 minutes. The Investigators are avoiding tilt test methods with provocative medications to avoid the issue of multiple causal factors. At 10 minutes and 30 minutes following onset of tilt (or at the onset of severe presyncope or hypotension [systolic BP <70 mmHg]), venous fractionated catecholamines will be sampled. The study will be terminated if the subject develops syncope or at the completion of the protocol.

3.10. Assessment of Central Volume Changes with Upright Posture: Segmental bioelectrical impedance (BEI) will measure fluid shifts through the study to determine central volume changes with upright posture and in response to changing levels of CO2. The fluid content in the upper torso (chest), the lower torso (abdominal), thigh, and calf will be assessed. BEI is measured by passing a small current between electrodes and measuring the impedance with voltage-sensing electrodes to determine fluid content in four regions of the body . Body segment volume is inversely proportional to electrical resistance (V~1/R), so an increase in resistance reflects a loss of body fluid.

3.11. Questionnaires: A brief online questionnaire will be administered to the patients to get a metric of their health-related quality of life (RAND-36), and anxiety and depression symptoms (HADS). This will be administered through RedCap Survey.

ELIGIBILITY:
Inclusion Criteria:

(A) ≥1 syncopal spells in the year preceding enrolment (B) ≥-2 points on the Calgary Syncope Symptom Score( Accurate Calculation for Diagnosis of Vasovagal Syncope) (C) Age ≥18 years with informed consent

Exclusion Criteria:

1. other causes of syncope, such as ventricular tachycardia, complete heart block, orthostatic hypotension or hypersensitive carotid sinus syndrome
2. an inability to give informed consent
3. important valvular, coronary, myocardial or conduction abnormality or significant arrhythmia
4. hypertrophic cardiomyopathy
5. a permanent pacemaker
6. a seizure disorder
7. hypertension defined as >160/90 mm Hg
8. pregnancy
9. lactating women
10. glaucoma
11. medications with known effects on BP
12. Known hypersensitivity to ondansetron and related medications
13. other factors which, in the investigator's opinion, would prevent the subject from completing the protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to syncope or presyncope | 1 hour

SECONDARY OUTCOMES:
stroke volume | 1 hour
cardiac output | 1 hour
  Heart Rate * Stroke volume, and it will be measured using Beat -To Beat BP measurement and HR measurement
catecholamine levels | 1 hour
Hospital Anxiety and Depression Scale (HADS) | Within 12 months period of the study
  The total score is out of 42, (21 per subscale). Scores are derived by summing responses for each of the two subscales or for the scale as a whole Higher scores indicate greater levels of anxiety or depression. The total HADS score may be regarded as a global measure of psychological distress
RAND-36 | Within 12 months period of the study
  The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. Aggregate scores are compiled as a percentage of the total points possible, using the RAND scoring table
systemic vascular resistance | 1 hour
  it will be measured using Beat -To Beat BP measurement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No